CLINICAL TRIAL: NCT01086683
Title: Rehabilitation of Cancer Survivors in Denmark: A Randomized Controlled Trial on the Effect of a Multi-focused Psychosocial Rehabilitation Course
Brief Title: Rehabilitation of Cancer Survivors in Denmark: The Effect of a Psychosocial Rehabilitation Course
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Danish Cancer Society (Other)
Collaborators: University Hospital Århus, Department of Surgery (Unknown); University Hospital Århus, Urology Department (Unknown); Randers Regional Hospital (Other); Regional Hospital Hørsholm, Department of Breast Surgery (Unknown)
Responsible Party: Professor Christoffer Johansen, MD, PhD, DMSc, Department of Psychosocial Cancer Research, Institute of Cancer Epidemiology, The Danish Cancer Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 225 06 001
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2010-03-15 (Estimated); Status verified 2010-03

CONDITIONS: Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms
Keywords: neoplasms; rehabilitation; intervention; quality of life; lifestyle
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: Psychosocial rehabilitation course
- Control group (No Intervention): Wait list control group: The control group received usual care including clinical control visits but no systematic rehabilitation activities.

INTERVENTIONS:
Behavioral: Psychosocial rehabilitation course — Groups of 20 cancer survivors participated in a 6-day multi-focused, psychosocial intervention at the Dallund rehabilitation centre. The overall aim was to strengthen each individual's physical, psychological and social functioning. Sharing experiences with other cancer patients and experiencing peer-support was a central issue. The retreat combined lectures, discussions and patient group work on themes such as the treatment of cancer, psychological reactions, spirituality, sexuality and lifestyle. Participants were involved in physical activities, and the daily menu represented a healthy diet. The course was conducted by a multi-disciplinary team. Each participant produced a personal, specific 'action plan', which was intended to serve as a 'booster' after returning to daily life.
  Arms: Intervention group

SUMMARY:
This randomized study evaluates the effect of a multi-focused, psychosocial 6-day residential rehabilitation course at a Danish rehabilitation centre for cancer survivors. The investigators hypothesize that individuals in the intervention group will experience better psychosocial well-being and more adaptive health behaviour changes as compared to individuals in the control group.

DETAILED DESCRIPTION:
Worldwide, the number of cancer survivors is increasing. In the Danish population of 5.4 million people, more than 300 000 are cancer survivors. Given the range of physical, psychological and social late effects of cancer and its primary treatment many survivors need tailored rehabilitation interventions. This randomized study evaluates the effect of a multi-focused, psychosocial 6-day residential rehabilitation course at the Dallund Rehabilitation Centre in Denmark. We hypothesize that individuals in the intervention group will experience better psychosocial well-being and more adaptive health behaviour changes as compared to individuals in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of breast, colorectal or prostate cancer
* Completion of primary treatment
* Ability to participate physically in the activities offered in the intervention

Exclusion Criteria:

* Acute need for treatment
* Terminal cancer phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2004-05; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
psychosocial well-being (as assessed by the EORTC-QLQ C30 Quality of life core questionnaire by the European Organization of Research and Treatment in Cancer (EORTC-QLQ C30) and the Profile of Mood States Short form (POMS-SF) | baseline, 1 month follow-up, 6 month follow-up, 12 month follow-up
  self-report questionnaire

SECONDARY OUTCOMES:
health behaviours: physical activity, diet, tobacco and alcohol consumption, use of health services | baseline, 1 month, 6 month, 12 month follow-up
  self-report questionnaire
self-rated health | baseline, 1 month, 6 month, 12 month follow-up
  self-report item
self-efficacy as measured with the General Self-Efficacy Scale (GSE) | baseline, 1 month, 6 month, 12 month follow-up
  self-report questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Johansen, MD, PhD, Principal Investigator — Department of Psychosocial Cancer Research, Institute of Cancer Epidemiology and National Centre for Cancer Rehabilitation Research, University of Southern Denmark
Locations (1):
- Department of Psychosocial Cancer Research, Copenhagen, Denmark

REFERENCES:
- [Derived] Ibfelt E, Rottmann N, Kjaer T, Hoybye MT, Ross L, Frederiksen K, Johansen C, Dalton SO. No change in health behavior, BMI or self-rated health after a psychosocial cancer rehabilitation: Results of a randomized trial. Acta Oncol. 2011 Feb;50(2):289-98. doi: 10.3109/0284186X.2010.531761. PMID 21231790